CLINICAL TRIAL: NCT01272791
Title: A Randomized, Open-Label, Phase 2 Trial of Gemcitabine With or Without Bavituximab in Patients With Previously Untreated Stage IV Pancreatic Cancer
Brief Title: Trial of Gemcitabine With or Without Bavituximab in Patients With Previously Untreated Stage IV Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PPHM 1002
Record Dates: First submitted 2011-01-03; First posted 2011-01-10 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: metastatic stage IV pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — bavituximab; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gemcitabine, bavituximab (Experimental): Gemcitabine will be administered on Days 1, 8, 15 of each 28-day (4 weeks) cycle until disease progression or unacceptable toxicities. Patients randomized to receive bavituximab will receive 3 mg/kg weekly (in addition to gemcitabine) until disease progression or unacceptable toxicities
  Interventions: Biological: bavituximab
- Gemcitabine (Active Comparator): Patients randomized to Gemcitabine (1000 mg/m2) will be given on Days 1, 8 and 15 of each 28 day cycle (4 weeks) until disease progression or unacceptable toxicities.
  Interventions: Drug: Gemcitabine

INTERVENTIONS:
Biological: bavituximab — Patients who qualify for enrollment into the study will be randomized in a 1:1 ratio to receive study treatment of gemcitabine alone or gemcitabine with weekly 3 mg/kg bavituximab. Treatment for each patient will begin on Study Day 1. Gemcitabine (1000 mg/m2) will be given on Days 1, 8 and 15 of each 28 day cycle (4 weeks) until disease progression or unacceptable toxicities. Patients randomized to receive bavituximab will be treated weekly beginning on Day 1 of each cycle. Study visits are scheduled to occur every 7 (± 2) days for bavituximab administration (for patients randomized to receive bavituximab); gemcitabine administration will occur every 7 (± 2) days for the first 3 weeks of each 4-week cycle
  Other Names: Gemzar
  Arms: Gemcitabine, bavituximab
Drug: Gemcitabine — Gemcitabine (1000 mg/m2) will be given on Days 1, 8 and 15 of each 28 day cycle (4 weeks) until disease progression or unacceptable toxicities
  Other Names: Gemzar
  Arms: Gemcitabine

SUMMARY:
The primary objective of this study is to compare the overall survival of patients with stage IV pancreatic cancer treated with gemcitabine alone or gemcitabine with bavituximab.

DETAILED DESCRIPTION:
This is prospective, randomized, open-label, multicenter, phase 2 study of gemcitabine with or without bavituximab in patients with previously untreated stage IV pancreatic cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent has been obtained.
* Adults of 18 years of age or older with a life expectancy of at least 3 months.
* Patients with histologically or cytologically documented stage IV ductal adenocarcinoma of the pancreas.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate hematologic function (ANC ≥ 1,500 cells/µL; hemoglobin ≥ 9 g/dL, platelets ≥ 100,000/µL).
* Adequate renal function (serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 60 mL/min).
* Adequate hepatic function (bilirubin ≤ 1.5 x ULN, ALT ≤ 3 x ULN, AST ≤ 3 x ULN); ALT and AST may be <5 x ULN if due to liver metastases.
* PT/INR ≤ 1.5 × ULN.
* aPTT ≤ 1.5 × ULN.
* Female patients must have a negative urine or serum pregnancy test at screening (pregnancy test not required for patients with bilateral oophorectomy and/or hysterectomy or for those patients who are > 1 year postmenopausal).
* All patients of reproductive potential must agree to use an approved form of contraception (as determined by the investigator).

Exclusion Criteria:

* Neuroendocrine tumors (carcinoid, islet cell cancer) of the pancreas.
* NYHA Class III or IV, cardiac function, myocardial infarction within 6 months prior to Day 1, unstable arrhythmia or symptomatic peripheral arterial vascular disease.
* Known brain, leptomeningeal or epidural metastases.
* Radiation therapy within 7 days of Study Day 1, lack of recovery from previous therapeutic radiation, or planned radiation therapy during the study period.
* Previously received any systemic treatment for pancreatic cancer, including prior neoadjuvant or adjuvant chemotherapy for lower stage disease.
* Previously malignancies, except for adequately treated non-melanoma skin cancer, in situ cancer, or other cancer from which the subject has been disease-free for at least 5 years.
* Severe chronic obstructive or other pulmonary disease with hypoxemia.
* Major surgery, other than diagnostic surgery, within 4 weeks prior to Day 1, without complete recovery.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Ongoing therapy with oral or parenteral anticoagulants; patients on low-dose anticoagulants to maintain patency of lines are eligible.
* Venous thromboembolic events (e.g. deep vein thrombosis or pulmonary embolism) within 6 months of screening.
* QTC interval of >470 ms on screening.
* Long QT syndrome or family history of sudden cardiac death in young family members.
* Subjects who participated in an investigational drug or device study within 28 days prior to study entry.
* Known active infection with HIV, hepatitis B, or hepatitis C.
* Females who are pregnant or breast-feeding.
* Concomitant disease or condition that could interfere with the conduct of the study, or that would, in the opinion of the investigator, pose an unacceptable risk to the subject in this study.
* Unwillingness or inability to comply with the study protocol for any reason.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Overall survival of patients with stage IV pancreatic cancer treated with gemcitabine alone or gemcitabine with bavituximab. | One year
  To compare the overall survival of patients with stage IV pancreatic cancer treated with gemcitabine alone or gemcitabine with bavituximab.

SECONDARY OUTCOMES:
Progression-free survival of patients with stage IV pancreatic cancer treated with gemcitabine alone or gemcitabine with bavituximab. | One year
  To compare the progression-free survival of patients with stage IV pancreatic cancer treated with gemcitabine alone or gemcitabine with bavituximab.
Determine overall response rate (ORR) | One year
  To determine the overall response rate [complete response (CR) and partial response (PR)] in stage IV pancreatic cancer treated with gemcitabine alone or gemcitabine with bavituximab.
Duration of response (DR) | One year
  To determine the duration of response (DR) in each treatment arm.
Determine the frequency of 25% or greater reduction in CA 19-9 in patients with baseline CA 19-9>=2 time the upper limit of normal (ULN) at screening | One year
  To determine the frequency of 25% or greater reduction in CA 19-9 in patients with baseline CA 19-9>=2 time the upper limit of normal (ULN) at screening in each treatment arm
Safety | One year
  To evaluate safety by treatment arm

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sklenar, Study Chair — Peregrine Pharmaceuticals
Locations (19):
- United States (15):
  - Ironwood Cancer & Research Centers, Chandler, Arizona
  - Moores UCSD Cancer Center, La Jolla, California
  - Lynn Cancer Institute, Boca Raton, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - The Cancer Center at DeKalb Medical, Decatur, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Nancy N. and J.C. Lewis Cancer & Research Pavilion at St. Joseph's/Candler, Savannah, Georgia
  - Joliet Oncology-Hematology Associates, Ltd., Joliet, Illinois
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Arena Oncology Associates, PC, Lake Success, New York
  - Leo W. Jenkins Cancer Center - East Carolina University, Greenville, North Carolina
  - St. Luke's Cancer Center, Bethlehem, Pennsylvania
  - Vasicek Cancer Center at Scott & White Memorial Hospital, Temple, Texas
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
- Ukraine (4):
  - Municipal Institution "Cherkasy Regional Oncology Dispensary" of Cherkasy Regional Council, Cherkasy
  - City Multi-field Clinical Hospital, Dnipropetrovsk
  - Municipal Institution of Health Care "Kharkiv Regional Clinical Oncology Center", Kharkiv
  - Kyiv City Oncology Center, Kyiv